CLINICAL TRIAL: NCT05668806
Title: Study of Real-world Evidence in Patients Treated With Cerviron Vaginal Ovules in the Treatment of Cervical Lesions of Various Etiology
Brief Title: RWE Study in the Treatment of Cervical Lesions of Various Etiology
Status: Completed | Type: Observational
Sponsor: Perfect Care Distribution (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Other Study IDs: CYRONRW/02/2022
Record Dates: First submitted 2022-11-18; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Cervical Lesion; Vaginal Bleeding
Keywords: cervical ectropion; vaginal discharge; cervix lesion
MeSH Terms: conditions — Uterine Hemorrhage; Vaginal Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cerviron — Cerviron® is an invasive medical device of short-term use classified under annex VIII of the European Regulation 2017/745 as class IIb according to Rule 21 (devices composed of substances or of combinations of substances to be introduced into the human body via a body orifice or applied to the skin and absorbed by or locally dispersed in the human body). Cerviron® has a complex composition consisting of three topical pharmaceutical products - hexylresorcinol, collagen and bismuth subgallate - and four phytotherapeutic extracts - Calendula officinalis, Hydrastis canadensis, Thymus vulgaris extract and Curcuma longa. The Instructions for use specify its field of use as adjuvant in the treatment of acute and chronic vulvovaginitis of mechanical etiology, caused by changes of vaginal pH and changes of the vaginal flora and of cervical lesions of mechanical origin.

SUMMARY:
The aim of the study was to assess the post-market performance and tolerability of Cerviron® ovules in the treatment and management of cervical lesions of different etiologies. The study included clinical data related to aspect of lesions performed during routine colposcopy exams, the degree of re-epithelialization of the cervical mucosa, vaginal pH, pain level, and vaginal bleeding level.

DETAILED DESCRIPTION:
This study is an observational, post-marketing study conducted between May-July 2021.

The aim of the study was to assess the post-market performance and tolerability of Cerviron® ovules in the treatment and management of cervical lesions of different etiologies.

The secondary objective of this clinical investigation is the assessment of performance of the medical device by clinical exam and patients' degree of satisfaction related to the use of the medical device.

The study population included 345 participants aged 20-70 years with either a cervical lesion under treatment or with recent surgical removal of a cervical lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clearly diagnosed non-infectious gynecological disease and patients with traumatic or surgical lesions.
* Patients with either of the following medical history: trauma of the cervix, pain, bleeding after sexual intercourse, postpartum injuries or postoperative cervical lesions.

Exclusion Criteria:

* Patients with cervical cancer.
* Patients with vulvar cancer

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are taking oral contraceptives often have cervical ectopy (cervical erosions).
Study Population: Women aged above 18 years with a clearly diagnosed non-infectious gynecological disease and patients with traumatic or surgical lesions.
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of treatment-related adverse events in subjects participating in the clinical investigation | 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Clinical Performance assessed by the investigator | 3 months
  An assessment of the cervical lesions by gynecological examination (visual evaluation)
Patient Satisfaction | 3 months
  An assessment on a 5-point Likert scale to evaluate the degree of satisfaction after the treatment. The scale rates satisfaction from Very satisfied (maximum) to Very unsatisfied (minimum).

CONTACTS AND LOCATIONS:
Overall Officials: Ema Peta, Study Director — Perfect Care Distribution
Locations (15):
- Romania (15):
  - Spitalul Clinic Dr. Ion Cantacuzino Bucharest, Bucharest
  - Med Life Humanitas Cluj-Napoca, Cluj-Napoca
  - Cabinet Medical - Dr. Saleh K. Majed, Craiova
  - Cabinet Medical - Dr. Surpanelu Oana, Iași
  - MediBlue, Iași
  - Clinica Natisan Pitesti, Piteşti
  - Cabinet Dr. Rădulescu G. Mihaela Elena, Râmnicu Vâlcea
  - Ramnicu Valcea, Râmnicu Vâlcea
  - Cabinet Ginecologic Dr. Popescu Sibiu, Sibiu
  - Clinica iMED, Sibiu
  - Pan Medical Sibiu, Sibiu
  - Bradmed SRL, Târgu Jiu
  - Cabinet Dr. Ioana Trotea Targu Jiu, Târgu Jiu
  - Clinica Medicala Dr. Cioata Ionel Trifon, Timișoara
  - Spitalul Judetean de Urgenta Tulcea, Tulcea

REFERENCES:
- [Derived] Petre I, Sirbu DT, Petrita R, Toma AD, Peta E, Dimcevici-Poesina F. Real-world study of Cerviron(R) vaginal ovules in the treatment of cervical lesions of various etiologies. Biomed Rep. 2023 Jul 7;19(2):54. doi: 10.3892/br.2023.1618. eCollection 2023 Aug. PMID 37546352